CLINICAL TRIAL: NCT02234882
Title: Effect of BMS-663068 on the Pharmacokinetics of Rosuvastatin
Brief Title: Study on Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 206276; AI438-048 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Rosuvastatin Calcium; fostemsavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin and BMS-663068 (Experimental): Treatment A: Rosuvastatin, single dose (SD) Treatment B: BMS-663068 administered on specified days Treatment C: Combination BMS-663068 and Rosuvastatin administered on specified days
  Interventions: Drug: Rosuvastatin; Drug: BMS-663068

INTERVENTIONS:
Drug: Rosuvastatin
Drug: BMS-663068

SUMMARY:
The purpose of this study is to assess the effect of the coadministration of multiple doses of BMS-663068 on the systemic exposure of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form

   * Signed written informed consent must be obtained from the subjects in accordance with requirements of the study center's IRB or IEC before the initiation of any protocol-required procedures.
2. Target Population

   * Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination findings, vital sign measurements, 12-lead ECG measurements, and clinical laboratory test results.
3. Age and Reproductive Status

   * Men and women of non-childbearing potential, ages 18 to 50 years, inclusive. Women must have documented proof that they are not of childbearing potential. Women must not be breastfeeding.
   * Males who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s).

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding
* Any significant acute or chronic medical illness
* History of rhabdomyolysis or biliary disorders, including Gilbert's disease or Dubin-Johnson disease
* Smokers (those who currently smoke, as well as those who have stopped smoking less than 6 months prior to the start of study drug administration)
* Alcohol intake exceeding 2 standard drinks per days; however, no alcohol is allowed 1 week prior to the start of study drug administration and for the duration of the study
* Any other sound medical, psychiatric, and/or social reason as determined by the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of rosuvastatin | Days 1 through 13
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) of rosuvastatin | Days 1 through 13

SECONDARY OUTCOMES:
Trough blood samples of BMS-626529 concentration | Days 7 through 13
Safety assessments based on review of adverse events, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests. | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: ViiV Clinical Trials, MD, Study Director — ViiV Healthcare